CLINICAL TRIAL: NCT00812747
Title: Surgical Wound Infections After Vascular Surgery: Prospective Multicenter Trial
Status: Completed | Type: Observational
Sponsor: North Karelia Central Hospital (Other)
Collaborators: Kuopio University Hospital (Other); South Carelia Central Hospital (Other); South Savo Hospital District (Other)
Responsible Party: MD Johanna Turtiainen, north karelia central hospital, clinic of surgery
Other Study IDs: NKCH-Surg-002
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Surgical Wound Infection
Keywords: surgical wound infection; risk factor
MeSH Terms: conditions — Surgical Wound Infection | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: observation

INTERVENTIONS:
Other: observation

SUMMARY:
The purpose of this multicentre prospective trial is to determine the incidence and risk factors for surgical wound infections. Also the investigators will evaluate consequences of wound infections to the patients, and extra costs caused by wound infections.

ELIGIBILITY:
Inclusion Criteria:

* non-emergency infrarenal aortic or lower limb arterial surgery

Exclusion Criteria:

* patient's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent non-emergency infrarenal aortic or lower limb arterial surgery between June 2007 and January 2008 were enrolled to this study.
Sampling Method: Non-Probability Sample
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
wound infection incidence

CONTACTS AND LOCATIONS:
Locations (1):
- North Karelia Central Hospital, Joensuu, Finland